CLINICAL TRIAL: NCT02461108
Title: Nudging Nutrition: Evaluating the Impact of Monetary Incentives and Environmental Cues on Food Choices
Brief Title: Nudging Nutrition With Monetary Incentives Environmental Cues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Ohio State University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 1110002491; 1RC1HD063370-01 (NIH)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Food Labeling; Health Behavior; Diet
Keywords: Public policy; Food choice; Nutrition labeling; Fat tax; Vegetable subsidy; Behavioral economics; Health behavior
MeSH Terms: conditions — Obesity; Health Behavior | interventions — Taxes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Price difference (Experimental): Introduce a 10% price difference between foods labeled as nutritious and foods labeled as less nutritious and frame the price difference as either a Subsidy, Tax, or combination of a Tax and Subsidy.
  Interventions: Behavioral: Subsidy; Behavioral: Tax; Behavioral: Tax and subsidy
- No price difference (No Intervention): No price difference between nutritious and less nutritious foods.

INTERVENTIONS:
Behavioral: Subsidy — Frame the price difference as a 10% subsidy on nutritious food items.
  Arms: Price difference
Behavioral: Tax — Frame the price difference as a 10% tax on less nutritious food items.
  Arms: Price difference
Behavioral: Tax and subsidy — Frame the price difference as a 5% tax on less nutritious food items and a 5% subsidy on nutritious food items, creating a 10% relative price difference between the types of foods.
  Arms: Price difference

SUMMARY:
The investigators hypothesize that monetary incentives and messaging, such as making nutritious foods relatively less expensive than less nutritious foods and framing the price difference in a positive or negative way, will influence purchasing behavior of households.

DETAILED DESCRIPTION:
In this study, 239 loyalty card shoppers were recruited at Hannaford grocery stores to participate in a study in which a 10% price difference between nutritious and less nutritious foods was introduced. and then framed as a subsidy, tax, or a combination of a tax and subsidy. To determine whether or not the framing of the price difference influenced purchasing behavior, the difference was framed as a subsidy on nutritious foods, a tax on less nutritious foods, and a combination of a tax and subsidy on less nutritious and nutritious foods, respectively. The purpose of this study was to examine the general impact of this price difference on purchases of nutritious and less nutritious foods, and whether or not the framing of the price difference had a differential effect on behavior.

ELIGIBILITY:
Inclusion Criteria:

* Loyalty card shoppers at Hannaford grocery stores

Exclusion Criteria:

* No children in household
* Less than 75% of food purchases made at Hannaford grocery stores

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in expenditures on nutritious and less nutritious foods | 8 months
  Item level transaction data were collected for each participant between mid-July 2010 and mid-March 2011. These data included expenditures on all items purchased in the store. Average weekly expenditures were generated and reported in Aug 2011.

SECONDARY OUTCOMES:
Change in quantities purchased of nutritious and less nutritious foods | 8 months
  Item level transaction data were collected for each participant between mid-July 2010 and mid-March 2011. These data included quantities of all items purchased in the store. Average weekly quantities purchased were generated and reported in Aug 2011.
Change in expenditures on nutritious and less nutritious foods in specific food categories. | 8 months
  Item level transaction data were collected for each participant between mid-July 2010 and mid-March 2011. These data included expenditures on all items purchased in the store, as well as the specific product type. With this information, product groupings can be created, such as for dairy, candy, and fresh produce. Average weekly expenditures for these groupings were generated and reported in July 2012.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Wansink, PhD, Study Director — Cornell University; David Just, PhD, Principal Investigator — Cornell University
Locations (1):
- New York City School District, New York, New York, United States

REFERENCES:
- [Result] Pope L, Hanks AS, Just DR, Wansink B. New Year's res-illusions: food shopping in the new year competes with healthy intentions. PLoS One. 2014 Dec 16;9(12):e110561. doi: 10.1371/journal.pone.0110561. eCollection 2014. PMID 25514158